CLINICAL TRIAL: NCT04594356
Title: Assessment of Netosis During COVID-19, Under Treatment With Anakinra, an Interleukin-1 Receptor Antagonist
Acronym: NET_COV
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: NET_COV
Record Dates: First submitted 2020-10-19; First posted 2020-10-20 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19 infection: As part of this research, existing clinical data of patients infected with COVID-19 is collected from the patients' computerized medical records.
  During the hospitalization of the patients, in addition to the clinical and laboratory data collected, the dosage of IL-6, apparently playing a central role in the worsening of the symptoms of COVID-19, was performed. The remainder of the contents of the tube used to perform this assay will allow further research by assaying the DNA-myeloperoxidase (DNA-MPO) complexes. These complexes reflect a phenomenon called "netosis," most likely involved in the widespread inflammation that patients have suffered from.

SUMMARY:
During their activation in response to an infectious stimulus or during chronic inflammatory processes, blood and tissue neutrophils modify their functional phenotype and produce numerous toxic mediators. In particular, they rapidly release chromatin filaments covered with numerous granular and cytoplasmic components called "Neutrophil Extracellular Traps" (NETs). This phenomenon, called netosis, has been implicated in many diseases, in particular in viral infections during which this response can be useful for the anti-infectious response at the initial phase, then deleterious when it becomes toxic. for the tissue environment. This has been shown in particular during post-pneumonia acute respiratory distress syndrome.

The intensity of netosis is therefore an early factor in activating neutrophils and inflammation. Given the major biological signs of inflammation observed in patients with COVID-19 as soon as they enter the hospital [C-Reactive protein (CRP), Interleukin-6 (IL-6), D-dimers, etc.), it seems particularly interesting to better document this inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients hospitalized within the Paris Saint-Joseph Hospital Group for whom the diagnosis of COVID-19 has been established on the basis of a PCR positive for SARS-CoV 19 using a nasal swab and/or a typical chest CT scan
* Patients with a severe or aggravating form of COVID-19, based on an oxygen saturation ≤93% under 6 l/min of nasal oxygen or a saturation ≤93% under 4 l/min oxygen with a decrease in saturation of at least 3% during the last 24 hours, in ambient air
* Patients treated with Anakinra
* Patients for whom IL-6 assays have been performed
* French speaking patients

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized within the Paris Saint-Joseph Hospital Group for whom the diagnosis of COVID-19 has been established on the basis of a PCR positive for SARS-CoV 19 using a nasal swab and or a typical chest CT scan, with a severe or aggravating form of COVID-19, based on an oxygen saturation ≤93% under 6 l / min of nasal oxygen or a saturation ≤93% under 4 l/min oxygen with a decrease in saturation of at least 3% during the last 24 hours, in ambient air
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the netosis process | Day 1
  This outcome corresponds to the of the determination of DNA-myeloperoxidase complexes (DNA-MPO).

SECONDARY OUTCOMES:
Evaluation of the netosis process at day 3 | Day 3
  This outcome corresponds to the of the determination of DNA-myeloperoxidase complexes (DNA-MPO).
Link between this marker (DNA-MPO) and the clinical course of patients | Day 3
  This outcome is to evaluate the clinical course of patients according to the DNA-MPO marker.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles HAYEM, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - CHU Bichat Claude Bernard, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Twaddell SH, Baines KJ, Grainge C, Gibson PG. The Emerging Role of Neutrophil Extracellular Traps in Respiratory Disease. Chest. 2019 Oct;156(4):774-782. doi: 10.1016/j.chest.2019.06.012. Epub 2019 Jun 29. PMID 31265835
- [Background] Granger V, Peyneau M, Chollet-Martin S, de Chaisemartin L. Neutrophil Extracellular Traps in Autoimmunity and Allergy: Immune Complexes at Work. Front Immunol. 2019 Dec 3;10:2824. doi: 10.3389/fimmu.2019.02824. eCollection 2019. PMID 31849989
- [Background] Bendib I, de Chaisemartin L, Granger V, Schlemmer F, Maitre B, Hue S, Surenaud M, Beldi-Ferchiou A, Carteaux G, Razazi K, Chollet-Martin S, Mekontso Dessap A, de Prost N. Neutrophil Extracellular Traps Are Elevated in Patients with Pneumonia-related Acute Respiratory Distress Syndrome. Anesthesiology. 2019 Apr;130(4):581-591. doi: 10.1097/ALN.0000000000002619. PMID 30676417
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Correction to: Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 Jun;46(6):1294-1297. doi: 10.1007/s00134-020-06028-z. PMID 32253449
- [Background] Sarzi-Puttini P, Giorgi V, Sirotti S, Marotto D, Ardizzone S, Rizzardini G, Antinori S, Galli M. COVID-19, cytokines and immunosuppression: what can we learn from severe acute respiratory syndrome? Clin Exp Rheumatol. 2020 Mar-Apr;38(2):337-342. doi: 10.55563/clinexprheumatol/xcdary. Epub 2020 Mar 22. PMID 32202240
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Kupferschmidt K, Cohen J. Race to find COVID-19 treatments accelerates. Science. 2020 Mar 27;367(6485):1412-1413. doi: 10.1126/science.367.6485.1412. No abstract available. PMID 32217705
- [Background] Mahase E. Covid-19: what treatments are being investigated? BMJ. 2020 Mar 26;368:m1252. doi: 10.1136/bmj.m1252. No abstract available. PMID 32217607
- [Background] Li G, De Clercq E. Therapeutic options for the 2019 novel coronavirus (2019-nCoV). Nat Rev Drug Discov. 2020 Mar;19(3):149-150. doi: 10.1038/d41573-020-00016-0. No abstract available. PMID 32127666
- [Result] Granger V, Fels A, Huet T, Laplanche JL, Laplanche S, Chatellier G, Beaussier H, Chollet-Martin S, de Chaisemartin L, Hayem G. Circulating IL-6 but not neutrophil extracellular traps levels can predict anakinra effectiveness in patients with severe COVID-19. J Leukoc Biol. 2022 Dec;112(6):1365-1367. doi: 10.1002/JLB.4LT0122-018RR. Epub 2022 Jun 15. PMID 35704508